CLINICAL TRIAL: NCT04068155
Title: A Safety and Effectiveness Study of Intratumoral Diffusing Alpha Radiation Emitters for the Treatment of Malignant Cutaneous Tumors
Brief Title: Alpha Radiation Emitters Device for the Treatment of of Malignant Cutaneous Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-MCT-00
Record Dates: First submitted 2019-08-19; First posted 2019-08-28 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Skin Cancer; Cutaneous Tumor; Cutaneous Metastasis
Keywords: Squamous Cell Carcinoma; Basal Cell Carcinoma; Skin Cancer; Skin Metastasis; Superficial Sarcoma; Alpha Radiation; Cutaneous Lesion; Brachytherapy; Radiotherapy; Lentigo maligna melanoma; Carcinosarcom; scalp cancer; Lip cancer; Eyelid cancer; SCC
MeSH Terms: conditions — Skin Neoplasms; Carcinoma, Squamous Cell; Carcinoma, Basal Cell; Lip Neoplasms; Eyelid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DaRT Seeds Intratumoral Diffusing alpha-emitters (Experimental): An intratumoral insertion of securely fixed seeds loaded with Radium-224. The seeds release by recoil short-lived alpha-emitting atoms into the tumor.
  Interventions: Device: DaRT- Diffusing Alpha-emitters Radiation Therapy

INTERVENTIONS:
Device: DaRT- Diffusing Alpha-emitters Radiation Therapy — Seed(s) loaded with Radium-224 for local intratumoral irradiation with the destructive power of alpha particles

SUMMARY:
A unique approach for cancer treatment employing intratumoral diffusing alpha radiation emitter device for Malignant Cutaneous Tumors

DETAILED DESCRIPTION:
This will be a prospective, open label, single arm, multi- center study, assessing the safety and effectiveness of diffusing alpha emitters radiation therapy (DaRT) delivered through radioactive seeds inserted into the tumor.

This approach combines the advantages of local intratumoral irradiation of the tumor, as used in conventional brachytherapy, with the power of the alpha radiation emitting atoms, that will be introduced in quantities considerably lower than radiation therapy already used in patients.

Cutaneous lesions with histopathological confirmation of malignancy will be treated using DaRT seeds.

Reduction in tumor size 9-11 weeks following DaRT insertion will be assessed. Safety will be assessed by the frequency, severity and causality of all Adverse Events (AE).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histopathological confirmation of newly diagnosed (Cohort A) or locally recurrent (Cohort B) malignant cutaneous lesions of the following histopathologies:

  * SCC
  * BCC
  * Lentigo maligna melanoma (Dubreuilh melanoma)
  * Carcinosarcoma
* Acceptable tumor locations include the following:

  * Skin (facial, scalp, extremities, torso)
  * Lips
  * Eyelids
* Subjects with a tumor size ≤ 7 centimeters in the longest diameter.
* Target lesion technically amenable for full tumor coverage with the Alpha DaRT seeds.
* Measurable disease according to RECIST v1.1.
* Subjects over 18 years old.
* Subjects' ECOG Performance Status Scale is < 2.
* Subjects' life expectancy is more than 6 months.
* Platelet count ≥100,000/mm3.
* International normalized ratio of prothrombin time ≤1.8.
* Women of childbearing potential (WOCBP) will have evidence of negative pregnancy test.
* Subjects are willing to sign an informed consent form

Exclusion Criteria:

* Subject has a tumor with histology of one of the following:

  * Keratoacanthoma
  * Merkel cell carcinoma
  * Sarcoma other than carcinosarcoma
* Metastatic disease (according to the TNM staging system - M1 patients are excluded)
* Patients with significant comorbidities that the treating physician deems may conflict with the endpoints of the study (e.g., poorly controlled autoimmune diseases, vasculitis, etc.).
* Patients undergoing systemic immunosuppressive therapy excepting intermittent, brief use of systemic corticosteroids.
* Volunteers participating in another interventional study in the past 30 days which might conflict with the endpoints of this study or the evaluation of response or toxicity of DaRT.
* High probability of protocol non-compliance (in opinion of investigator).
* Subjects not willing to sign an informed consent.
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
The objective response rate to DaRT treatment | up to 9-11 weeks
  Assessment of tumor response rate using the Response Evaluation Criteria in Solid Tumors (RECIST) (Version 1.1)

SECONDARY OUTCOMES:
Tumor volume | up to 9-11 weeks
  Assessment of the reduction in tumor volume based on imaging tests
DaRT seeds placement | Day of DaRT insertion procedure
  Assessment of the DaRT seed placement by localization of the DaRT seed in the tumor using CT imaging
Change in quality of life as assessed by the Skindex-16 questionnaire | up to 9-11 weeks
  Assessment of patient reported health-related Quality of Life (QoL) outcomes using the Skindex-16 questionnaire
Disease-Free Survival (DFS) rate | up to 24 months
  Assessment of Disease-Free Survival
Change in quality of life as assessed by the Skin Cancer Index (SCI) questionnaire | up to 9-11 weeks
  Assessment of patient reported health-related Quality of Life (QoL) outcomes using the Skin Cancer Index (SCI) questionnaire.

OTHER OUTCOMES:
Adverse Events | up to 24 months
  Assessment of the frequency, severity and causality of adverse events related and not related to the DaRT treatment. Adverse events will be assessed and graded according to Common Terminology and Criteria for adverse events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Pascal POMMIER, Principal Investigator — Centre Leon Berard; Pr Jean Michel HANNOUN LEVI, Principal Investigator — Antoine Lacassagne Cancer Center; Dr Camille VERRY, Principal Investigator — University Hospital, Grenoble
Locations (2):
- France (2):
  - CHU Grenoble Alpes, Grenoble
  - Centre Léon Bérard, Lyon

IPD SHARING:
Plan to Share IPD: No